CLINICAL TRIAL: NCT01616095
Title: The Effect of a Long-Term Growth Hormone Supplementation on the Whole-Body Metabolic Characteristics and Adipose Tissue Phenotype in Growth Hormone Deficient Adults: the 5-yr Follow-up
Brief Title: Effects of Growth Hormone Supplementation to Adults With Growth Hormone Deficient on Metabolism and Adipose Tissue Molecular Phenotype
Acronym: GHAT
Status: Completed | Type: Observational
Sponsor: Slovak Academy of Sciences (Other Government)
Collaborators: PFIZER, Bratislava, Slovakia (Unknown)
Responsible Party: Principal Investigator, Jozef Ukropec, PhD, Slovak Academy of Sciences
Other Study IDs: GH GIIR - 2011
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth hormone deficiency; hrGH therapy; metabolic health; adipose tissue metabolism; adipose tissue inflammation; adipokines
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — plasma 2.5 ml, serum 5 ml, adipose tissue 300 mg taken by the percutaneous biopsy of abdominal subcutaneous adipose tissue, in local anaesthesia.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Adults with Growth Hormone Deficiency: if multiple hormonal deficiences exist, long term adequate supplementation is provided and tightly monitored.
- Healthy Controls: matched for BMI, age, and gender

SUMMARY:
This study is designed as a follow up study to that performed in 2005.

In the Baseline study (2005) extensive clinical whole body metabolic phenotyping was combined with in depth molecular and cellular biology analyses aimed at investigating the adipose tissue morphology as well as metabolic and inflammatory phenotypes in the adult GHD patients. Results published in (Ukropec et al., 2008)

In this study identical endpoints will be investigated with the same methodology and within the same population; in order to seek relevant answers to questions on how the 6-yrs of rhGH therapy affects the

* whole body insulin sensitivity
* energy expenditure
* body fat distribution
* hepatic and skeletal muscle lipid content;

as well as how it influences the adipose tissue

* endocrine,
* metabolic &
* inflammatory phenotypes.

The strength of the planned study lies in the extensive whole body and adipose tissue phenotyping before and after the 6-year rhGH replacement therapy, that allows to determine the long-term effects of rhGH replacement therapy in GHD adults.

Envisaged weakness is the limited size of the population; GHD adults (n=20); controls [age BMI and gender matched] (n=20). This, however, reflects [is limited by] the complexity of the study protocol as well as the stringency of the inclusion criteria.

The clinical data obtained by methods of - integrated physiology would provide an excellent interpretation background for molecular-genetic studies at the tissue (adipose tissue) and cellular (adipocytes) level. Integration of the two could bring a new quality in the investigators understanding of metabolic derangements present in GHD, and will allow extending the investigators knowledge on the mechanisms of the long-term rhGH-therapy-induced improvement on body composition, metabolic health and the cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

We will follow inclusion-exclusion criteria which are very much like those used in the pilot study performed in 2005.

* Briefly, duration of the GHD prior to entering the study should last for at least 3 years prior rhGH treatment starts. Age of individuals eligible to enter should be 20-50 years old. All patients and healthy control volunteers will provide the witnessed written informed consent before entry into the study.
* It has to be noted that differences in the etiology of GHD might influence several of the outcomes we plan to measure. Presence or absence of possible bias should therefore be excluded for each specific outcome prior further statistical data analysis. Individuals with different degree of pituitary deficiency will therefore be eligible to enter the study.
* Complex information on the adequacy of the hormone replacement therapy will be based on the serum levels of growth hormone, insulin-like growth factor 1, free thyroid hormone, testosterone/estradiol, urinary free cortisol FT4, and morning cortisol. Examination and laboratory testing relevant to this study will be performed within 6 months of entering the study. The 24-hour urinary free cortisol will only be determined in individuals hospitalized in a period of two month prior to the study entry.

Exclusion Criteria:

* None of the patients should receive lipid lowering treatment. Patients with malignant disease, diabetes mellitus, existing vascular disease and uncontrolled hypertension are not eligible to enter this study.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty growth hormone deficient adults, receiving supplementation with rhGH for 5 years (extensively examined in 2005-2006, prior to the start of rhGH therapy) and 20 age-, gender- and BMI- matched controls will enter the study. Both, GHD patients and controls will undergo an extensive clinical protocol, identical to that performed in 2005 (Ukropec et al., 2008a).
  The possibility of drop-out of patients needs to be taken into consideration. Possible lowering of the numbers of participants due to drop-out of individuals tested in the Baseline Study will be resolved by either (i) using biological material obtained in the Baseline Study which was originally not subjected to an extensive molecular genetic testing due to the limited capacity and high cost of these analyses and/or by (ii) recruiting necessary amount of new patients with history of 5 years rhGH therapy (initial examination is missing).
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Effects of GH therapy to GHD adults - the whole body level | 12 months
  to determine the effects of a long-term (6 years) growth hormone supplementation on the whole-body metabolic phenotype in adult GHD patients (namely (i) insulin sensitivity, (ii) energy expenditure, (iii) body fat distribution and (iv) bone mineral density, (v) glucose tolerance, (vi) hepatic and skeletal muscle lipid content as well as (vii) serum lipids and (viii) inflammatory markers in circulation.
GH therapy effects on the endocrine, metabolic & inflammatory properties of adipose tissue | 2 years
  to investigate the effects of long-term (5 years) growth hormone supplementation on the subcutaneous adipose tissue (i) endocrine, (ii) metabolic and (iii) inflammatory phenotype in adult GHD patients, by extensive profiling of adipose tissue protein & gene expression (protein antibody arrays & real-time PCR) which could identify potential molecular mechanisms associated with abdominal obesity and insulin resistance modulated by rhGH replacement therapy.

SECONDARY OUTCOMES:
comparison of GHD & control population | 2 years
  to compare the whole-body metabolic profile and subcutaneous adipose tissue phenotype of rhGH supplemented GHD adults with that of the healthy control group
Identification of the adiposity-associated parameters | 2 years
  to evaluate parameters associated primarily with adiposity which are largely independent on the severity of the GH deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Ukropec, PhD, Principal Investigator — Inst. Exp. Endocrinology SAS, Bratislava, Slovakia; Barbara Ukropcova, MD, PhD, Study Chair — Inst. Exp. Endocrinology SAS, Bratislava, Slovakia; Iwar Klimes, prof, MD, PhD, Study Director — Inst. Exp. Endocrinology SAS, Bratislava, Slovakia; Daniela Gasperikova, PhD, Study Chair — Inst. Exp. Endocrinology SAS, Bratislava, Slovakia; Juraj Payer, prof, MD, PhD, Study Chair — Dep. of Endocrinology, University Hospital, Comenius University, Bratislava; Martin Kuzma, MD, Study Chair — Dep. of Endocrinology, University Hospital, Comenius University, Bratislava; Mikulas Pura, MD, PhD, Study Chair — National Institute of Diabetology and Endocrinology, Lubochna, Slovakia; Peter Vanuga, MD, PhD, Study Chair — National Institute of Diabetology and Endocrinology, Lubochna, Slovakia; Miroslav Vlcek, MD, PhD, Study Chair — Inst Exp. Endocirnology SAS, Bratislava; Adela Penesova, MD, PhD, Study Chair — Inst Exp. Endocirnology SAS, Bratislava; Miroslav Balaz, Mgr., Study Chair — Inst Exp. Endocirnology SAS, Bratislava; Timea Kurdiova, Mgr., Study Chair — Inst Exp. Endocirnology SAS, Bratislava
Locations (3):
- Slovakia (3):
  - V th Internal Clinic, Univeristy Hospital Bratislava, Comenius University, Bratislava
  - Inst. Exp. Endocrinology Slovak Acad Sci, Bratislava
  - National Institute of Endocrinology and Diabetology, Ľubochňa

REFERENCES:
- [Background] Ukropec J, Penesova A, Skopkova M, Pura M, Vlcek M, Radikova Z, Imrich R, Ukropcova B, Tajtakova M, Koska J, Zorad S, Belan V, Vanuga P, Payer J, Eckel J, Klimes I, Gasperikova D. Adipokine protein expression pattern in growth hormone deficiency predisposes to the increased fat cell size and the whole body metabolic derangements. J Clin Endocrinol Metab. 2008 Jun;93(6):2255-62. doi: 10.1210/jc.2007-2188. Epub 2008 Mar 11. PMID 18334583
- See also: link to the website of the Institute of Experimental Endocrinology Slovak Academy of Sciences — http://www.endo.sav.sk/